CLINICAL TRIAL: NCT03952598
Title: Studying the Biology of Higher-Grade Transformation in IDH-mutant Gliomas Via Longitudinal Observation of Tumor Metabolic Reprogramming Using Non-invasive Metabolic Imaging
Brief Title: Studying the Biology of IDH-mutant Gliomas Via Longitudinal Observation of 2-hydroxyglutarate (2-HG) Using MR Spectroscopy
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study on hold pending possible updates with the team.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 190096; 19-C-0096
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Glioma; Gliomas; High Grade Glioma; Malignant Glioma; Low Grade Glioma
Keywords: Imaging; Higher-Grade Transformation; Biomarker for Cancer; High Grade Gliomas
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Arm 1 (Experimental): Monitoring of quantitative levels of 2-hydroxyglutarate (2-HG) via proton magnetic resonance spectroscopy (1H-MRS) -- THIS ARM IS NOW CLOSED
  Interventions: Device: 3T MRI scanner
- 2/Arm 2 (Experimental): Monitoring of quantitative levels of 2-hydroxyglutarate (2-HG) via proton magnetic resonance spectroscopy (1H-MRS) and HP 13C pyruvate MRSI
  Interventions: Device: 3T MRI scanner
- 3/Arms 3 (Experimental): Monitoring of quantitative levels of 2-hydroxyglutarate (2-HG) via proton magnetic resonance spectroscopy (1H-MRS)
  Interventions: Drug: HP 13C Pyruvate; Device: 3T MRI scanner

INTERVENTIONS:
Drug: HP 13C Pyruvate — Contrast agent used with magnetic resonance spectroscopic imaging (MRSI)
  Arms: 3/Arms 3
Device: 3T MRI scanner — Research proton MRS (1H-MRS) followed by DW-MRI

SUMMARY:
Background:

Glioma is a type of brain cancer. Some of these tumors have gene mutations. These mutations can cause a substance called 2-HG to build up in the brain. This makes the tumors more aggressive. Researchers want to better understand 2-HG buildup in the brain. They hope this can help them design better ways to test for gliomas.

Objective:

To monitor the level of 2-HG in the brains of people with gliomas that have mutations in the IDH1 or IDH2 genes.

Eligibility:

People ages 18 and older with gliomas with mutations in the IDH1 or IDH2 genes

Design:

Participants will be screened with:

Medical and cancer history

Physical exam

Reviews of their symptoms and ability to perform normal activities

Blood and urine tests

MRI scan

Samples of their tumor from a past surgery

Documentation of their diagnosis and mutation status

Participants will have an initial evaluation. This will include repeats of screening tests. It will also include:

Neurological exam

MRS and MRI scans of the brain: Participants will lie on a table that slides into a metal cylinder. A coil or soft padding will be placed around their head. They will have a contrast agent injected into a vein. Pictures will be taken of the brain.

Participants will have follow-up visits every 2-6 month for the rest of their life. Visits will include scans.

DETAILED DESCRIPTION:
Background:

* Glioma is the most common malignant brain tumor. Genes coding for isocitrate dehydrogenase (IDH), a metabolic enzyme, are frequently mutated in gliomas, particularly lower-grade gliomas (LGGs). IDH mutation causes a unique tumor biology, including the accumulation of 2-hydroxyglutarate (2-HG), an oncometabolite, which in turn causes genomic hypermethylation and tumorigenesis.
* Despite having a better prognosis compared to their IDH WT counterparts, IDH-mutant LGGs undergo a slow but unremitting higher-grade transformation (HT) and eventually become high grade gliomas (HGGs). A subset of patients with transformed HGGs develop a hypermutator phenotype (HMP), possibly related to previous treatment with alkylating agents. The timeline for the development of HT and HMP is unpredictable and there is no known way to prevent them from happening, largely due to a lack of understanding their biological mechanisms and lack of a non-invasive approach for potential early detection.
* Metabolic imaging, including proton magnetic resonance spectroscopy (MRS) and hyperpolarized (HP) 13C-Pyruvate MRSI, can safely detect the in vivo metabolic changes in humans.
* This clinical study will allow a longitudinal monitoring of participants with IDH-mutant gliomas for detection of disease progression, which is associated with metabolic alterations, provide an unprecedented opportunity for biopsy of the tumor for diagnostic confirmation and interrogation of the mechanisms of HT and HMP, and potentially providing a specific treatment approach for HMP which has been refractory to conventional brain tumor treatments.

Objective:

To detect and monitor the quantitative levels of 2-HG and lactate/pyruvate ratio longitudinally in participants with IDH-mutant gliomas via proton MRS and HP 13C pyruvate MRSI, respectively

Eligibility:

* Participant has glioma harboring IDH1 or IDH2 mutation confirmed by DNA sequencing.
* Age >=18 years, KPS >= 70%

Design:

* This is a prospective observational study. We will recruit up to 270 eligible participants in the next 5 years.
* The relationship between the occurrence of HT and the changes in 2-HG level and the ratio of lactate/pyruvate will be evaluated using the proportional hazard model with the latter as the time-dependent covariates.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically confirmed diffuse glioma with documented IDH1 or IDH2 mutation, confirmed by DNA sequencing the exception will be participants with brain lesions that are not safe for biopsy but clinically suspected to be diffuse glioma are allowed to enroll to the study to receive imaging study as part of the exploratory study
* Participants must have measurable disease.
* Age >=18 years. Tumor biology of IDH-mutant gliomas are different in pediatric tumors. Therefore, children will be excluded from the study.
* Karnofsky performance >= 70%.
* Participants must have documented normal kidney function as defined below:

Creatinine within normal institutional limits

OR

Creatinine clearance >60 mL/min/1.73 m2 for Participants with creatinine levels above institutional normal (Measured or calculated creatinine clearance

-Participants must have adequate liver function as defined below:

total bilirubin <=2x ULN (ULN 1.3 mg/dl) except for participants with Gilbert Syndrome

AST < 3x ULN (ULN 34U/L)

ALT < 3x ULN (ULN 55U/L)

-Ability of participants to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of this study, and that this is not a therapeutic clinical trial.

EXCLUSION CRITERIA:

* Participants who have contraindication to MRI examination, including, but not limited to, unable to receive gadolinium, medical instability, or any contraindication on MR Screening Form. Pregnant individuals are excluded because MRI contrast, planned to be used on this study, may be dangerous for the fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to using of MRI contrast, breastfeeding should be discontinued for 72 hours following study imaging.
* Participants weighing > 350 lbs. (weight limit for scanner table), or unable to fit within the imaging gantry
* Poorly controlled hypertension, with blood pressure >150/90 mmHg.
* Congestive heart failure with New York Heart Association (NYHA) status > 2.
* A medical history of clinically significant EKG abnormalities, including QT prolongation, a family history of prolonged QT interval syndrome, or myocardial infarction (MI) less than 1 year ago with ensuing unstable EKG.
* Ongoing acute or chronic pulmonary bronchospastic disease, including a history of chronic obstructive pulmonary disease or asthma with an exacerbation within the past year.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To monitor the quantitative levels of 2-hydroxyglutarate (2-HG) longitudinally in patients with IDH mutant gliomas via proton magnetic resonance spectroscopy (1H-MRS) | 5 years
  Changes in the level of 2-HG correlate with the occurrence of higher-grade transformation (HT) and/or development of hypermutator phenotype (HMP) in patients with IDH-mutant gliomas

SECONDARY OUTCOMES:
Determine the utility of 2-HG detection by 1H-MRS to predict higher-grade transformation (HT) and hypermutator phenotype (HMP) by correlating the 2-HG level with pathological diagnosis and tumor mutational load of the tumor tissue at time of rec... | at clinical disease recurrence
  Usefulness of 2-HG detection and its correlation with high grade transformation and HMP

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
BTRIS: All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@dbGaP: All large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: BTRIS: Clinical data available during the study and indefinitely.@@@@@@dbGaP: Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: BTRIS: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@dbGaP: Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0096.html